CLINICAL TRIAL: NCT04312113
Title: A Phase I Single Site Open Label Study of Intra-arterial Delivery of Mesenchymal Stem Cells for Luminal Ulcerative Colitis
Brief Title: Angiographic Delivery of AD-MSC for Ulcerative Colitis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William A. Faubion, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-000826
Record Dates: First submitted 2020-03-14; First posted 2020-03-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous mesenchymal stem cells (Experimental): Adipose derived, autologous mesenchymal stem cells (AD-MSCs) at a dose of 15 million or 30 million cells will be administered via intra-arterial delivery with interventional radiology to the inferior mesenteric artery in subjects with medically refractory ulcerative colitis.
  Interventions: Drug: Adipose derived, autologous mesenchymal stem cells

INTERVENTIONS:
Drug: Adipose derived, autologous mesenchymal stem cells — Fat tissue will be enzymatically treated and cells will be cultured until a sufficient number are obtained for the treatment protocol.
  Other Names: AD-MSC

SUMMARY:
Researchers are trying to determine the safety and feasibility of using an adipose derived mesenchymal stem cell (MSC) to treat people with Ulcerative Colitis.

DETAILED DESCRIPTION:
Participants will undergo screening for study, if eligible, participants will be dosed with 15 million or 30 million cells will be administered via IA delivery with interventional radiology. Participant study visits after study intervention includes visits on: Day 1, Week 1, Week 2, Week 8, Week 24, Week 52, and Week 104.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females 18-65 years of age.
* Moderate to Severe medically refractory inflammatory ulcerative colitis:

  * as defined by a an Adapted Mayo Score of 5to 9 points
  * including an endoscopic sub-score of 2 or 3
* Concurrent therapies with corticosteroids, 5-ASA drugs, thiopurines, MTX, antibiotics, anti-TNF, and anti-integrin therapy are permitted.
* To meet the definition of refractory UC, all patients must have failed at least 2 standard FDA approved medications for the treatment of UC

  * Current standard therapy includes 5-ASA products, thiopurines, anti-TNF therapy, ustekinemab, vedolizumab, and tofacitinib (i.e. all FDA approved therapies for UC).
  * Refractory and failure to response is defined as continued symptoms despite 12 weeks of therapy at FDA approved doses by product necessitating change in medical strategy or referral for colectomy.
* All patients should have undergone a colonoscopy in last 12 months to rule out malignant or premalignant condition
* Female subjects that are of child bearing potential must to agree to use effective contraception method(s) for the duration of the study
* Hemoglobin must be greater than 8
* INR must be less than 1.5
* Ability to comply with protocol
* Competent and able to provide written informed consent

Exclusion Criteria:

* Inability to give informed consent.
* Clinically significant medical conditions within the six months before administration of MSCs: e.g. myocardial infarction, active angina, congestive heart failure or other conditions that would, in the opinion of the investigators, compromise the safety of the patient.
* Specific exclusions; Known history of hepatitis B, C, or HIV
* Patients that have had a partial colectomy
* Patients that have underlying vasculitis or have been diagnosed with an underlying condition that predisposes to developing blood clots.
* History of cancer including melanoma (with the exception of localized skin cancers)
* Investigational drug within thirty (30) days of baseline
* History of clinically significant auto-immunity (other than UC) or any previous example of fat-directed autoimmunity. Note that auto-immmunity is defined as a systemic immune mediated disease for which the antigen is known or unknown. Autoimmune diseases other than UC are excluded. Extraintestinal manifestations of UC (specifically joint inflammation, eye inflammation, PSC, skin manifestations- i.e. pyoderma gangrenosum, erythema nodosum) will be allowable.
* Allergic to local anesthetics
* Pregnant patients or trying to become pregnant or breast feeding.
* Neoplasia of the colon and preoperative biopsy
* C. Difficile infection within 30 days of study injection
* Diagnosis of indeterminate colitis or suspicion of CD
* Subjects with fulminant colitis, toxic megacolon, with ostomy, or ileoanal pouch
* History or demonstration of pathology related to adipose tissue
* Any other indication determined by the PI to be counter indicated for participation on this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events | 24 months
  Evaluate safety by assessment of adverse events defined as worsening (change in nature, severity, or frequency of bowel movements, bleeding per rectum, or tenesmus) of UC present at the time of the study, intercurrent illnesses, abnormal laboratory values (this includes clinically significant shifts from baseline within the range of normal that the investigator considers to be clinically significant) or clinically significant abnormalities in physical examination, vital signs, weight, frequency of bloody stools or change in stools.

SECONDARY OUTCOMES:
Number of participants with mucosal healing | 6 months
  Mucosal appearance at endoscopy via Adapted Mayo Score (defined as score of 0 or 1)
Number of participants with clinical symptom response | 24 months
  To assess the clinical symptom response of luminal healing induced by the intra-arterial delivery of autologous AD-MSCs for the treatment of UC. Using the validated via Adapted Mayo Score (decrease from Baseline ≥ 2 points and ≥ 30%, including a decrease in rectal bleeding sub-score ≥ 1 or an absolute rectal bleeding sub-score ≤ 1)
Number of participants with improved healing on pathology | 24 months
  Histopathology: Improved healing on surgical pathology (colectomy specimen or post-intervention colonic biopsies) as compared to pre-operative endoscopic biopsies

CONTACTS AND LOCATIONS:
Overall Officials: William Faubion, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials